CLINICAL TRIAL: NCT04594473
Title: The Feasibility and Acceptability of a Comprehensive Oncology Rehabilitation and Exercise (CORE) Program Among Breast Cancer Survivors
Brief Title: A Comprehensive Oncology Rehabilitation and Exercise (CORE) Program Among Breast Cancer Survivors
Acronym: CORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adriana Coletta, Assistant Professor, Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00137018
Record Dates: First submitted 2020-10-12; First posted 2020-10-20 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Survivors; Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): Participants randomized to SOC will be instructed to continue their typical lifestyle activity.
- Comprehensive Oncology Rehabilitation and Exercise (CORE) Program (Experimental): Participants randomized to CORE will be instructed to follow the clinical algorithm for this study. An in-clinic assessment consisting of two questionnaires will be used to identify the appropriate pathway for triage. Participants will be triaged into one of three pathways: Physical Medicine & Rehabilitation, Personal Optimism With Exercise Recovery, or Exercise Self-Management.
  Interventions: Behavioral: Comprehensive Oncology Rehabilitation and Exercise (CORE) Program

INTERVENTIONS:
Behavioral: Comprehensive Oncology Rehabilitation and Exercise (CORE) Program — [see arm/group descriptions]
  Arms: Comprehensive Oncology Rehabilitation and Exercise (CORE) Program

SUMMARY:
The objective of this study is to demonstrate the feasibility and acceptability of the algorithm utilized within a cancer rehab program, named Comprehensive Oncology Rehabilitation and Exercise (CORE) program, among newly diagnosed stage I-III breast cancer survivors, providers, and clinic staff. Additionally, this study aims to generate preliminary estimates on the extent to which CORE, compared with standard of care (SOC), elicits engagement in exercise and impacts changes in physical function and quality of life within this population.

DETAILED DESCRIPTION:
Enrollment: The study team will recruit 72 newly diagnosed stage I-III breast cancer survivors to participate in a 24-week randomized controlled trial. Participants will be randomized to CORE or SOC in a 2:1 ratio, stratified by adherence to national physical activity guidelines.

Exercise Intervention: Participants randomized to standard of care will be instructed to continue their typical lifestyle activity. Participants randomized to CORE will complete an in-clinic assessment consisting of the PROMIS Physical Function and Godin surveys to identify the appropriate pathway for triage. Results from the questionnaires will be used to triage participants into one of three groups:

1. Physical Medicine & Rehabilitation (PM&R): This rehab service is aimed at improving complex and acute functional deficits. Participants with a T-score < 40 on PROMIS will be triaged to PM&R, regardless of current exercise engagement.
2. Personal Optimism With Exercise Recovery (POWER): POWER is our institution's exercise oncology program. POWER is aimed at improving mild functional deficits and physical deconditioning. Participants with a T-score of 40-50 on PROMIS who are not meeting activity guidelines, will be triaged to POWER. Participants with a T-score of ≥ 40 who are meeting activity guidelines, may choose to participate in POWER or be re-triaged to Exercise Self-Management.
3. Exercise Self-Management: This arm is aimed for participants who are fit and free of functional deficits and impaired physical conditioning. Participants with a T-score of ≥ 51 on PROMIS and currently meeting activity guidelines will be triaged to this group. They may choose to participate in POWER.

Assessments: Five assessment methods will be collected over three time points: (1) Post-Diagnosis/Pre-Surgery, (2) Post-Surgery, and (3) 24-weeks Post-Surgery.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage I-III breast cancer survivors who have plans to undergo breast cancer surgery

Exclusion Criteria:

* Stage I-III breast cancer survivors who had received neoadjuvant chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who complete in-clinic assessment | Measured at Post-Diagnosis/Pre-Surgery assessment
  Percentage of participants who complete the in-clinic assessment will be used to determine the feasibility of CORE. Clinic staff will ask the participant to complete the PROMIS and Godin surveys for triaging into the CORE algorithm. CORE will be considered feasible if ≥ 66% of participants complete the in-clinic assessment and are assigned to one of the three pathways in the algorithm.
Percentage of participants who complete their referral | Measured at Post-Diagnosis/Pre-Surgery assessment
  Percentage of participants who complete their referral to a service pathway will be used to determine the feasibility of CORE. If the participant is triaged into PM&R or POWER groups based on in-clinic assessment, provider will submit a referral in participant's electronic medical record. Once the referral is submitted, patient navigation staff will be notified and immediately reach out to the participant to schedule with the referred service. CORE will be considered feasible if ≥ 50% of those referred to a service pathway (PM&R or POWER) complete their referral.

SECONDARY OUTCOMES:
Percentage of themes identified from focus groups that contain positive feedback | Upon completion of 24-weeks post-surgery SOC visit for participants and about one year post-implementation (approximately 1 year into data collection)
  To determine the acceptability of CORE, the study team will conduct focus groups one year after implementation of CORE. Four focus groups will be conducted among participants in CORE, and one focus group will be conducted among providers and clinic staff.
Change in exercise engagement assessed via accelerometer | Measured one-week Post-Diagnosis/Pre-Surgery SOC visit, one-week Post-Surgery SOC visit, and one-week 24-Weeks Post-Surgery SOC visit
  Researchers will examine the extent to which CORE elicits exercise engagement before and after breast cancer surgery compared to standard of care. At each assessment visit, participants will be provided with an Actigraph GT9X Link tri-axial accelerometer to objectively assess exercise engagement, and will be instructed to wear the device for seven days following their assessment.
Change in exercise engagement assessed via modified Godin survey | Measured one-week Post-Diagnosis/Pre-Surgery SOC visit, one-week Post-Surgery SOC visit, and one-week 24-Weeks Post-Surgery SOC visit
  Researchers will examine the extent to which CORE elicits exercise engagement before and after breast cancer surgery compared to standard of care. At each assessment visit, participants will be asked to fill out the modified Godin survey that measures typical weekly frequency of engagement in strenuous, moderate, and mild aerobic exercise. The modified version also inquires about average length of time of aerobic exercise engagement and frequency of resistance exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Department of Health and Human Services. Physical Activity Guidelines for Americans, 2nd edition. Washing, DC: US. Department of Health and Human Services; 2018.
- [Background] Rothrock NE, Cook KF, O'Connor M, Cella D, Smith AW, Yount SE. Establishing clinically-relevant terms and severity thresholds for Patient-Reported Outcomes Measurement Information System(R) (PROMIS(R)) measures of physical function, cognitive function, and sleep disturbance in people with cancer using standard setting. Qual Life Res. 2019 Dec;28(12):3355-3362. doi: 10.1007/s11136-019-02261-2. Epub 2019 Aug 13. PMID 31410640
- [Derived] Simon LH, Saviers-Steiger C, Dunston ER, Galyean P, Kimball ER, Mendez J, Zickmund SL, Hansen PA, Ulrich CM, LaStayo PC, Steinberg D, Noren CS, Finch A, Seckinger L, Braun E, Chipman J, Brownson KE, Oza S, Coletta AM. Feasibility and acceptability of the Comprehensive Oncology Rehabilitation and Exercise (CORE) clinical workflow algorithm in patients with newly diagnosed stage I-III breast cancer who undergo surgery as first-line treatment. Cancer. 2025 May 1;131(9):e35798. doi: 10.1002/cncr.35798. PMID 40289623